CLINICAL TRIAL: NCT02409745
Title: The Effectiveness of Endometrial Injury in Different Phase of Menstrual Cycle:a Prospective Controlled Clinical Study
Brief Title: The Effectiveness of Endometrial Injury in IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RMCZZU-EEI
Record Dates: First submitted 2015-01-06; First posted 2015-04-07 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
Keywords: endometrial scratch; IVF; randomized controlled study; Prospective controlled trial; Different time to perform endometrial scratch; In vitro fertilization; embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Young age group-Luteal phase (Experimental): Endometrial injury in luteal phase (previous menstrual cycle) for patients undergoing Frozen thawed embryo transfer.
  Interventions: Procedure: endometrial scratch
- Young age group-Early follicular phase (Active Comparator): Endometrial injury in early follicular phase for patients undergoing Frozen thawed embryo transfer.
  Interventions: Procedure: endometrial scratch
- Advanced age group-Luteal phase (Experimental): Endometrial injury in luteal phase (previous menstrual cycle) for patients undergoing Frozen thawed embryo transfer.
  Interventions: Procedure: endometrial scratch
- Advanced age group-Early follicular phase (Active Comparator): Endometrial injury in early follicular phase for patients undergoing Frozen thawed embryo transfer.
  Interventions: Procedure: endometrial scratch

INTERVENTIONS:
Procedure: endometrial scratch — local injury to the endometrium by Pipelle
  Other Names: endometrial injury

SUMMARY:
Many studies have demonstrated that endometrial scratch significantly increase pregnancy rate in patients undergoing in vitro fertilization and embryo transfer. However, only a limited number of studies have been conducted in frozen thawed transfer (FET) cycle. Nowadays, in FET cycles, endometrial scratch is mainly performed on two different time points: 1) luteal phase in the previous cycle; 2)early follicular phase in the current cycle. However, few studies have compared the effectiveness of those two different endometrial scratch methods performed in different timing. The aim of this study is to find the best timing of endometrial scratch in FET cycles.

ELIGIBILITY:
Inclusion Criteria:

* To be aged younger than 40 years old;
* At least one period IVF-ET (fresh or thaw) has been done and not pregnant after at least one qualified blastocyst (more than 3BB) or two qualified embryos (more than II/6) have been transferred;
* There are qualified embryos thawed and the thaw-ET period will be taken.

Exclusion Criteria:

* Malformation of uterus: such as uterus uni-corns, uterus bi-corns, untreated uterus septus, etc.;
* History of endometrial diseases: such as intrauterine adhesion, uterine cavity tuberculosis, severe dysplasia of endometrium, etc.;
* Multiple myomata or endometrioma which causes uterus oppression;
* Multiple and recurrent endometrial polyps;
* Pelvic tuberculosis, endometriosis.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 35 days after embryo transfer
  See heart beat with ultrasonic exam.

SECONDARY OUTCOMES:
Ectopic pregnancy rate | 35 days after embryo transfer
  No sac can be seen inside uterine 35 days after embryo transfer, but with high hCG level

CONTACTS AND LOCATIONS:
Overall Officials: Yingpu Sun, MD,PhD, Study Chair — Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University
Locations (1):
- Reproductive Medical Center, 1st Affiliated hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Background] Yeung TW, Chai J, Li RH, Lee VC, Ho PC, Ng EH. The effect of endometrial injury on ongoing pregnancy rate in unselected subfertile women undergoing in vitro fertilization: a randomized controlled trial. Hum Reprod. 2014 Nov;29(11):2474-81. doi: 10.1093/humrep/deu213. Epub 2014 Sep 8. PMID 25205759
- [Background] Nastri CO, Lensen SF, Gibreel A, Raine-Fenning N, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2015 Mar 22;(3):CD009517. doi: 10.1002/14651858.CD009517.pub3. PMID 25803542
- [Background] Potdar N, Gelbaya T, Nardo LG. Endometrial injury to overcome recurrent embryo implantation failure: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Dec;25(6):561-71. doi: 10.1016/j.rbmo.2012.08.005. Epub 2012 Sep 12. PMID 23063812
- [Background] El-Toukhy T, Sunkara S, Khalaf Y. Local endometrial injury and IVF outcome: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Oct;25(4):345-54. doi: 10.1016/j.rbmo.2012.06.012. Epub 2012 Jun 26. PMID 22885017
- [Background] Dain L, Ojha K, Bider D, Levron J, Zinchenko V, Walster S, Dirnfeld M. Effect of local endometrial injury on pregnancy outcomes in ovum donation cycles. Fertil Steril. 2014 Oct;102(4):1048-54. doi: 10.1016/j.fertnstert.2014.06.044. Epub 2014 Jul 23. PMID 25064410